CLINICAL TRIAL: NCT01878227
Title: Randomized Head-to-Head Comparison of Coenzyme A Capsule and Fenofibrate for Safety and Efficacy On Patients With Hyperlipidemia: A Phase III, Multicenter, Double-blinded, Double Dummy Clinical Trial.
Brief Title: Comparison of Coenzyme A and Fenofibrate for Safety and Efficacy On Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jiangtao Lai, MD, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010MMXX2CoA007
Record Dates: First submitted 2013-06-10; First posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Hyperlipoproteinemia
MeSH Terms: conditions — Hyperlipoproteinemias | interventions — Coenzyme A; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coenzyme A 400mg (Experimental): Coenzyme A 400mg per day
  Interventions: Drug: Coenzyme A
- Fenofibrate 200mg (Active Comparator): Fenofibrate 200mg per day
  Interventions: Drug: Fenofibrate 200mg

INTERVENTIONS:
Drug: Coenzyme A — Coenzyme A 400mg per day
  Other Names: Coenzyme A group
  Arms: Coenzyme A 400mg
Drug: Fenofibrate 200mg — Fenofibrate 200mg per day
  Other Names: Fenofibrate group
  Arms: Fenofibrate 200mg

SUMMARY:
The purpose of this study is to compare the lipid lowering effects and clinical safety of a natural hypolipidemic compound, coenzyme A capsule with a marketed drug, fenofibrate, in Chinese patients with moderate dyslipidemia.

DETAILED DESCRIPTION:
Although lowering cholesterol and low-density lipoprotein-cholesterol (LDL-C) is the mainstay of medical therapy for cardiovascular event prevention, evidence from clinical trials supports a role for elevated triglyceride (TG) and low high-density lipoprotein cholesterol (HDL-C) concentrations in the residual cardiovascular risk on statin treatment. Fenofibrate is the most commonly used agent to control hypertriglyceridemia as monotherapy or combining with statin, which lowers TG and raises HDL-C through multifaceted mechanism by PPARα activation. However, safety of coadministration of statin with fenofibrate has been a great concern, especially drug-induced hepatotoxicity when they are combined used. Coenzyme A (CoA) functions as an acyl group carrier and assists in transferring fatty acids from the cytoplasm to mitochondria. It is also involved in the oxidation and catabolism of fatty acids. Animal studies have proved its lipid-lowering effects. In a previous multicenter study we conducted in 2008, it was found that oral CoA 400U/d effectively lowered serum TG levels in hypertriglyceridemia patients without increasing adverse effects when compared with placebo. So, the present study was performed to further investigate the lipid-lowing effects and safety of CoA capsule by comparing with fenofibrate.

ELIGIBILITY:
Inclusion Criteria:

* TG 2.3～6.5mmol/l
* 18-75 years of age

Exclusion Criteria:

* TC >7.0 mmol/l;
* Body Mass Index > 30 kg/m2
* drug induced secondary hypercholesterolemia (such as dibenzothiazine, contraceptive agent or adrenal cortex hormone)
* pregnancy
* acute coronary syndrome, acute myocardial infarction or undergone a revascularization procedure within 6 months
* acute liver disease or hepatic dysfunction, as determined by levels of alanine aminotransferase (ALT) or aspartate aminotransferase levels (AST) more than 3-fold the upper normal limit
* nephrotic syndrome or serum creatinine (Cr) (≥179 µmol/L) and creatine •phosphokinase (CK) more than 3-fold the upper normal limit
* primary hypothyroidism
* psychiatric patients
* poorly controlled hypertension, as indicated by a Systolic Blood Pressure >180 mmHg or Diastolic Blood Pressure >110 mmHg
* Type I diabetes mellitus（DM）, poorly controlled Type II DM (BS>11.0 mmol/L ) or Type II DM with LDL-C >2.6 mmol/L.
* using immunosuppressive drugs, prohibited medication or other lipid-lowing drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
serum triglyceride level | 10 months
  The primary efficacy variable was the percentage change in serum lipid level from baseline to 4 and 8 weeks of treatment.

SECONDARY OUTCOMES:
serum total cholesterol level | 10 months
  change from baseline to 4 and 8 weeks of treatment in serum total cholesterol level.
low-density lipoprotein cholesterol level | 10 months
  change from baseline to 4 and 8 weeks of treatment in serum low-density lipoprotein cholesterol level.
serum high-density lipoprotein cholesterol level | 10 months
  change from baseline to 4 and 8 weeks of treatment in serum high-density lipoprotein cholesterol level.

CONTACTS AND LOCATIONS:
Overall Officials: Junzhu Chen, Study Chair — Zhejiang University
Locations (1):
- 1st Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China